CLINICAL TRIAL: NCT04665973
Title: Effect of a Brief Therapeutic Patient Education Session on Physical Activity in Patients at the Onset of Cancer Therapy: A Randomized Controlled Trial
Brief Title: Effect of an Oral Therapeutic Patient Education Session on Physical Activity in Patients With Cancer
Acronym: ETAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ETAP
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cancer
Keywords: Therapeutic Patient Education; Physical Activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral semi-structured interview (Experimental): The oral semi-structured interview uses the principles of motivational interviewing (partnership with the patient, no judgment, altruism, evocation) and follow the content of the booklet used in the control group.
  Interventions: Behavioral: Therapeutic patient education : oral semi-structured interview
- Booklet (Active Comparator): The information booklet was designed by the physiotherapists at Cliniques universitaires Saint-Luc and is specifically dedicated to raise patient's awareness about the benefits of physical activity (PA) in the context of cancer.
  Interventions: Behavioral: Therapeutic patient education : booklet (passive)

INTERVENTIONS:
Behavioral: Therapeutic patient education : oral semi-structured interview — The physiotherapist discusses and goes through each page of the booklet and involves the patient as much as possible. He demonstrates the exercises proposed in the booklet and then ask the patient to perform them in front of him. The physiotherapist tries to identify the patient's needs and suggests different ways to ensure that the patient has different opportunities to maintain the best possible level of PA
  Arms: Oral semi-structured interview
Behavioral: Therapeutic patient education : booklet (passive) — The booklet (11 pages): explains why it is important to maintain a good level of PA as part of cancer treatment and reviews the most common side effects of cancer therapy and the relative importance of PA in combating these effects (pages 2-3) ; defines PA, its modalities and possible security precautions (pages 4-5), suggests exercises to be performed oneself and a target intensity to be reached (pages 6-8), provides a roadmap to be completed oneself (pages 9-10), and outlines procedures for joining an exercise medicine group (page 11).
  Arms: Booklet

SUMMARY:
Despite significant evolution of cancer therapies from the early 20th century, these therapies are still associated with toxic effects that negatively impact the patient's performance status, quality of life and survival. The role of physical activity to counteract these side effects is acknowledged. However, cancer patients are often misinformed about the potential benefits of physical therapy during cancer therapy. In this context, the role of therapeutic patient education seems essential.

Because of lack of time, therapeutic patient education (TPE) is often provided via an information booklet. However, the investigators assume that a face-to-face interview results in a greater impact on patient's behavior change (the level of physical activity during cancer therapy, in our case). This research project is designed to challenge this hypothesis. The investigators hypothesize that a brief oral educational session of 30 minutes provided at the very beginning of cancer therapy will enhance the physical activity level of our patients for at least 6 months, i.e. during their cancer therapy.

DETAILED DESCRIPTION:
The investigators aim to compare the effects of two forms of TPE on the patient's PA level. In one of the two forms, TPE is delivered using an information booklet accompanied with a semi-structured oral interview (intervention group), whereas in the other form TPE is only delivered via the booklet (control group). The investigators hypothesize that the brief oral educational session of 30 minutes provided at the very beginning of cancer therapy will enhance the PA level of our patients for at least 6 months, i.e. during their cancer therapy.

The study is designed as a double-blind randomized controlled trial. The primary outcome is the evolution in each group of the PA level (via the international physical activity questionnaire (IPAQ) - long form) between the start of cancer therapy and 6-month follow-up.

Eligible patients will be randomly assigned either to the intervention group (TPE includes the information booklet + the semi-structured oral intervention provided by a physiotherapist) or to the control group (TPE will consist only in the information booklet). Patients and assessors will be blinded.

The relative efficacy of these 2 treatment arms will be evaluated at baseline, after 3 months at a visit for a follow-up medical consultation set by the oncologist, and after 6 months at a second follow-up consultation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 84 years
* Suffering from a first cancer, with the exception of the following cancers in the patient's history (provided that they have been successfully treated):

  * non-melanoma skin cancer,
  * carcinoma in situ of the uterine cervix
  * ductal carcinoma in situ.
* Preserved performance status (ECOG scale ≤ 1),
* Starting one of the following systemic cancer therapies:

  * chemotherapy,
  * immunotherapy,
  * targeted therapies,
* Able to understand and read French
* Life expectancy of at least 1 year

Exclusion Criteria:

* Poor cognitive function (Mini-Mental State Examination ≤ 24/30)
* Having a recurrence of cancer, with the exception of the following cancers in the patient's history (provided that they have been successfully treated):

  * non-melanoma skin cancer,
  * carcinoma in situ of the uterine cervix,
  * ductal carcinoma in situ.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Changes in PA level | At baseline and 6 months (at the occasion of a second follow-up visit set with the oncologist) after the start of the cancer therapy
  The PA level will be estimated in MET/h/week via the International Physical Activity Questionnaire (long form) validated in French in subjects aged 18-84 years.
  The questionnaire classifies the subject according to 3 activity levels: inactive, moderate, high

SECONDARY OUTCOMES:
Changes in PA level | At baseline and 3 months (at the occasion of a first follow-up visit set with the oncologist) after the start of the cancer therapy
  The PA level will be estimated in MET/h/week via the International Physical Activity Questionnaire (long form) validated in French in subjects aged 18-84 years.
  The questionnaire classifies the subject according to 3 activity levels: inactive, moderate, high
Changes in BMI | At baseline, 3 months and 6 months after the start of the cancer therapy
  Body mass index (BMI) is measured as weight (kg) divided by height is meters squared (m²)
Changes in fatigue | At baseline, 3 months and 6 months after the start of the cancer therapy
  Fatigue is measured via the Functional Assessment of Chronic Illness Therapy - Fatigue scale (FACIT-F).
  The scale is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function.
  The total score range from 0 to 160. The lower the score, the higher the fatigue.
Changes in quality of life | At baseline, 3 months and 6 months after the start of the cancer therapy
  Quality of life is measured via the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30).
  The QLQ-C30 is composed of both multi-item scales and single-item measures. There are 30 items. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All single-item measures range in score from 0 to 100.
  A high score for a functional scale represents a high / healthy level of functioning, A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems.
Changes in exercise capacity | At baseline, 3 months and 6 months after the start of the cancer therapy
  Exercise capacity is measured via the 1-minute sit-to-stand test
Changes in handgrip strength test | At baseline, 3 months and 6 months after the start of the cancer therapy
  Handgrip strength test is measured via the JAMAR dynamometer
Number of steps | At 3 months and 6 months after the start of the cancer therapy
  The number of steps taken weekly via an application (ITO) downloaded on the patient's phone
Number of patients entering a group of exercise medicine | At 6 months after the start of the cancer therapy
  The proportion of patient who started a program of exercise medicine will be calculated in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium